CLINICAL TRIAL: NCT04664556
Title: Population-based Nationwide Study on Invasive Pneumococcal Infections Among Children (0-18 Years) in France
Brief Title: Invasive Pneumococcal Disease Study
Status: Recruiting | Type: Observational
Sponsor: Association Clinique Thérapeutique Infantile du val de Marne (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: IPD
Record Dates: First submitted 2020-12-07; First posted 2020-12-11 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Pneumococcal Infections; Pneumococcal Conjugate Vaccine; Antibiotic Treatment; Mortality
MeSH Terms: conditions — Pneumococcal Infections | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort of invasive pneumococcal disease in children
  Interventions: Other: observational study

INTERVENTIONS:
Other: observational study — observational study

SUMMARY:
After 7 then 13 valent pneumococcal conjugate vaccine implementation in France in children, we will evaluate the impact of this vaccination on invasive pneumococcal disease (IPD). We will describe the clinical characteristics of IPD, pneumococcus serotyping, underlying conditions and vaccination status.

ELIGIBILITY:
Inclusion Criteria:

* Isolate of Streptococcus pneumoniae from at least one blood culture, or pleural fluid, or joint fluid, or cerebrospinal fluid or other normally sterile body site, or if there is a positive blood PCR.

Exclusion Criteria:

* Pneumococcal strain not transmetted to National Reference Center for Pneumococci or to Regional Pneumococci Observatory

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with invasive pneumococcal disease for whom the pneumococcal strain is sent to the National reference Center for Pneumococci for serotyping
Sampling Method: Non-Probability Sample
Enrollment: 1369 (Estimated)
Dates: Start 2010-12-13 (Actual); Primary Completion 2030-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Severity of invasive pneumococcal disease | before hospital discharge
  Number of severe cases according to age and pneumococcal serotypes distribution

SECONDARY OUTCOMES:
Impact of vaccines | before hospital discharge
  Number of invasive pneumococcal disease according to vaccine serotypes

CONTACTS AND LOCATIONS:
Overall Officials: Levy Corinne, Study Director — Association Clinique Thérapeutique Infantile du val de Marne; Cohen Robert, Principal Investigator — Association Clinique Thérapeutique Infantile du val de Marne
Locations (1):
- ACTIV, Créteil, France

IPD SHARING:
Plan to Share IPD: Undecided